CLINICAL TRIAL: NCT05239520
Title: Understanding Control and Mechanisms of Shoulder Instability in Patients With Facioscapulohumeral Muscular Dystrophy (FSHD)
Brief Title: Understanding Control and Mechanisms of Shoulder Instability in FSHD
Status: Completed | Type: Observational
Sponsor: University of Liverpool (Other)
Collaborators: Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government); Bournemouth University (Other); Keele University (Other)
Responsible Party: Sponsor
Other Study IDs: UoL001656; RPG185 (Other Grant/Funding Number: The Orthopaedic Institute Ltd); Robert Jones & Agnes Hunt site (Other: RL1 811)
Record Dates: First submitted 2022-01-27; First posted 2022-02-15 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Shoulder Pain; Neuromuscular Diseases; Shoulder Injuries; Facio-Scapulo-Humeral Dystrophy; Upper Extremity Problem
Keywords: Biomechanics; Human movement analysis; Electromyography; Ultrasound
MeSH Terms: conditions — Shoulder Pain; Neuromuscular Diseases; Shoulder Injuries; Muscular Dystrophy, Facioscapulohumeral | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People affected by FSHD: Participants with a diagnosis of FSHD. 3D movement analysis session including surface electromyography and Ultrasound.
  Interventions: Other: 3D movement analysis with surface electromyography and ultrasound
- Age matched control group: Participants without a diagnosis of FSHD. 3D movement analysis session including surface electromyography and Ultrasound
  Interventions: Other: 3D movement analysis with surface electromyography and ultrasound

INTERVENTIONS:
Other: 3D movement analysis with surface electromyography and ultrasound — Single measurement session of 3D movement analysis with surface electromyography for upper limb movements and ultrasound measurements of upper muscles

SUMMARY:
The aim of this study is to identify factors for shoulder instability in people with Facioscapulohumeral dystrophy (FSHD). FSHD is a non-life limiting condition with symptoms presenting in the second decade of life (Evangelista et al., 2016). Between 2500 to 3000 people are diagnosed with FSHD in the UK and it is the third most common dystrophy. The overall prevalence is 1: 20,000 and on average 52 people are newly diagnosed with FSHD each year (Emery, 1991; Padberg et al., 1995; UK, 2020) As the disease progresses, patients lose the ability to adequately control muscles around the shoulder girdle, possibly contributing to the development of shoulder instability i.e. partial or complete dislocation of the shoulder joint (Bergsma, Cup, Geurts, & De Groot, 2015; Bergsma, Cup, Janssen, Geurts, & de Groot, 2017; Mul et al., 2016). Loss of control around the shoulder is also thought to contribute to pain and a reduced capacity to perform tasks above shoulder height. Additionally, the development of fatigue and chronic pain further limit patient's abilities and engagement with rehabilitation.

If we better understand the mechanisms associated with instability, we can better target physiotherapy interventions to improve rehabilitation. If we identify specific patterns of activity associated with instability, these could be addressed through personalised and improved exercise prescription and rehabilitation. Additionally, we may identify causes of instability for which physiotherapy or exercise programmes may not be appropriate, therefore ensuring patients are referred to the correct service in a timely manner, improving patient outcomes and allocating resources more appropriately.

DETAILED DESCRIPTION:
Shoulder instability in Facioscapulohumeral dystrophy (FSHD) is a significant problem, with over 80% of patients reporting that it affects their ability to perform activities of daily living (Faux-Nightingale , 2021). The underlying mechanisms of shoulder instability in FSHD are not well understood. It is thought that instability at the shoulder subsequently contributes to the development of shoulder pain and progressive loss of function, particularly during tasks performed above head height. Despite a large proportion of patients reporting shoulder instability that affects function, only 50% report engaging in some form of upper limb rehabilitation (Faux-Nightingale , 2021).

Both surgical and nonsurgical interventions are based on a current understanding of the associated mechanisms that may include muscle wasting, weakness, changes to the structure of the muscle tissue or inappropriate muscle coordination (Bergsma et al., 2014). As there is no cure for FSHD, rehabilitation is fundamental in the management of the condition. Overall, rehabilitation strategies are aimed at maintaining existing levels of function, avoiding complications associated with progression of the disease and targeting mechanisms associated with the development of instability. e.g. exercises to improve co-ordination of the shoulder muscles if the source of instability is dysfunctional muscle control.

Rehabilitation in patients with FSHD is complex and it is therefore important that rehabilitation is appropriately targeted. There is limited evidence to support the effectiveness of existing rehabilitation strategies in FSHD. In order for rehabilitation to be appropriately allocated disease mechanisms should be understood. Existing mechanisms of shoulder instability in FSHD are not well understood and may explain why more than 50% of patients are not engaging in any form of upper limb rehabilitation.

Shoulder stability results from complex mechanisms comprising of finely balanced forces in ligaments, muscles and joint surfaces (Ameln, Chadwick, Blana, & Murgia, 2019). Currently, we are unable to capture this complexity to quantify instability during dynamic upper limb tasks performed during clinical assessment and rehabilitation (Marchi, Blana, & Chadwick, 2014). Biomechanical or mathematical modelling of this complex structure can help to understand the mechanisms associated with instability and predict outcomes for surgical and non-surgical interventions (Arnold, Liu, Ounpuu, Swartz, & Delp, 2006; Delp et al., 2007; Laracca, Stewart, Postans, & Roberts, 2014). Loading on internal structures that cannot be measured can also be estimated by this approach.

This project is therefore a fundamental step, in the development of biomechanical models which can ultimately be used to further our understanding of the shoulder, specifically behaviour of the articulating bony surfaces and muscle forces. In this application we hope to identify mechanisms for shoulder instability which may help better inform rehabilitation and surgical decision making in the management of FSHD.

ELIGIBILITY:
People affected by FSHD

Inclusion Criteria:

Stratified groups

* Able to lift arms above shoulder height (n=3)
* Unable to lift arms above shoulder height (n=2)
* Post Scapulothoracic shoulder arthrodesis (n=2)
* Diagnosed with FSHD
* Aged 18 years and older

Exclusion Criteria:

* Recent trauma to the shoulder within the last 3 months on the arm being assessed that has not resolved
* Recent surgery to the thorax or upper limb in the last 6 months
* Previous history of fracture to the shoulder joint being assessed
* Co-existing neurological pathologies or additional musculoskeletal injuries to the upper limb being assessed

Age Matched Controls

Inclusion Criteria

- People aged 18 years and older

Exclusion Criteria:

* Any previous presentation to a health care professional with a diagnosis of shoulder instability
* Previous shoulder injury within the last 3 months on the arm being assessed that has not resolved
* Any co-existing neurological pathologies or deficits
* Any previous surgical intervention on the arm being assessed
* Currently undergoing or awaiting medical management, diagnostic investigations or rehabilitation on the arm being assessed

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will consist of people aged 18 years of age and older. The two groups will include people with (people affected by FSHD) and without FSHD (age matched controls).
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2022-10-21 (Actual)

PRIMARY OUTCOMES:
Kinematic features of movement: joint angles (degrees) | Day 1
  Range of movement values and associated derivatives will be reported for the associated movement tasks.
Kinematic features of movement: displacement (mm) | Day 1
  Displacement values and associated derivatives will be reported for associated movement tasks.
Kinetic variables related to the movement tasks: Force (Nm) | Day 1
  Force values for the strength testing, joint contact and muscle force values will be reported for associated movement tasks.
Muscle activity patterns related to the movement tasks: Surface electromyography (mv) | Day 1
  Muscle activity patterns related to the movement tasks will be reported for associated movement tasks.
Ultrasound imaging: Muscle architecture parameters (mm) | Day 1
  Muscle architecture parameters where possible (Muscle thickness)

CONTACTS AND LOCATIONS:
Locations (1):
- Robert Jones & Agnes Hunt Orthopaedic Hospital, Oswestry, Gobowen, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The anonymised final trial dataset and anonymised 3D movement data files will be stored on the University of Liverpool data repository. The anonymised dataset associated with the University of Liverpool data repository will be assigned a Digital object identifier and will be openly available.
Supporting Information: Study Protocol
URL: http://datacat.liverpool.ac.uk/